CLINICAL TRIAL: NCT06778135
Title: Neocortical Microarchitecture of Executive Function Using Large-scale Intracranial Electrophysiology
Brief Title: Neocortical Microarchitecture of Executive Function
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 23-1858; R61DC021924 (NIH)
Record Dates: First submitted 2025-01-10; First posted 2025-01-16 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Implanted (Experimental)
  Interventions: Procedure: Temporary implatation of large-scale intracranial electrode.; Device: brain electrode

INTERVENTIONS:
Procedure: Temporary implatation of large-scale intracranial electrode. — The Neuropixels probe (imec, Leuven, Belgium) is a new high resolution multi electrode technology that uses custom 130-nm complementary metal-oxide-semiconductor fabrication with high surface area but low-impedance titanium nitride recordings to produce high site count devices with extreme electrode density in a small package.
Device: brain electrode — Show that Neuropixels can safely and effectively record from large populations of neurons.

SUMMARY:
This study is being done to the determine the ability and utility of using the Neuropixels probes in the human brain. A Neuropixels probe will be inserted into and removed from the brain of awake human patients who are undergoing awake Deep Brain Stimulation (DBS) surgery.

DETAILED DESCRIPTION:
This project aims to use Neuropixels probes to record hundreds of neurons during awake human intracranial surgeries. Using this probe, we will take advantage of access to a key area in the network involved in executive function, the middle frontal gyrus of the dorsal lateral Pre Frontal Cortex (approximately the mid portion of dlPFC, part of Brodmann area 9/46), to test emerging concepts that cognitive flexibility so crucial to human EF is encoded in neural population geometry and layer-specific interactions.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Parkinson's disease and refractory to medications requiring deep brain stimulation
2. Aged 45-85
3. Able to provide informed consent
4. Normal neuropsychiatric evaluation that includes tests of executive function demonstrating no greater than mild impairments, within expectation for Parkinson's disease.
5. Medically able to undergo deep brain stimulation surgery as evaluated by study neurosurgeon.
6. Surgical plan includes an entry point that can safely be placed in the dorsal lateral PFC.
7. Able to tolerate awake deep brain stimulation surgery with a plan for the case to be done awake.
8. Able to tolerate 25 additional minutes of awake surgery.
9. Able to participate and comply with tasks adequately, including instructions provided in English.

Exclusion Criteria:

1. Moderate, or severe cognitive impairment as determined by a licensed neuropsychologist during routine neuropsychological evaluation.
2. Inability to tolerate awake surgery as determined by the treating neurologist and study neurosurgeon.
3. Inability to safely access the dorsal lateral prefrontal cortex for an entry location.
4. Moderate or severe cognitive impairment or executive function deficits as determined by neuropsychological testing.
5. Evidence of a clinically significant abnormality on preoperative imaging.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Measure the neural population representations of task parameters along, and within, the cortical layers. | 20 minutes

SECONDARY OUTCOMES:
Measure the neural population dimensionality in response to changing task parameters | 20 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado, Aurora, Colorado, United States